CLINICAL TRIAL: NCT05073783
Title: Multi-Centre, Non-Interventional, Double Cohort Study to Assess the Safety of Myozyme® and of Aldurazyme® in Real-World Home Infusion Setting
Brief Title: A Study to Assess the Safety of Myozyme® and of Aldurazyme® in Male and Female Participants of Any Age Group With Pompe Disease or With Mucopolysaccharidosis Type I (MPS I) in a Home-care Setting
Acronym: HomERT
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17128; U1111-1266-7312 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-09-16; First posted 2021-10-11 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Pompe Disease; Mucopolysaccharidosis Type I (MPS I)
MeSH Terms: conditions — Glycogen Storage Disease Type II; Mucopolysaccharidosis I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Pompe disease patients receiving Myozyme® (alglucosidase alfa) in a home-care setting.
- Cohort B: MPS I patients receiving Aldurazyme® (laronidase) in a home-care setting.

SUMMARY:
Primary objective:

To obtain data pertaining to the safety and tolerability of alglucosidase alfa and laronidase treatments administered in a home-care infusion setting.

Secondary objectives:

* To evaluate personal satisfaction of both cohorts of patients treated in a home-care infusion setting.
* To evaluate the infusion compliance in both cohorts of patients treated in a home-care infusion setting.

DETAILED DESCRIPTION:
Prospective observation duration for each patient: at least 12 months (from enrollment)

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent obtained prior to being enrolled into the study and prior to starting any data collection. Consent of a legally authorized guardian is required for legally minor patients as defined by local regulation. If the patient is legally minor, signed written consent shall be obtained from parent(s)/legal guardian and assent obtained from the patient, if applicable.
* Pompe disease patients with confirmed acid alpha-glucosidase (GAA) enzyme deficiency treated with Myozyme® in home infusion setting according to authorized clinical practice and the approved risk management plan document (Cohort A) or
* MPS I patients with confirmed deficiency of the lysosomal enzyme, alpha-L-iduronidase treated with Aldurazyme® in home infusion setting according to authorized clinical practice and the approved risk management plan document (Cohort B).

Exclusion Criteria:

* Participation in another clinical trial with any investigational agent within the 12 weeks preceding enrolment.
* Any condition (e.g. medical concern) which, in the opinion of the Investigator, would make the participant unsuitable for the study.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pompe disease patients with confirmed GAA enzyme deficiency treated with Myozyme® in home infusion setting according to authorized clinical practice and the approved risk management plan document (Cohort A) or MPS I patients with confirmed deficiency of the lysosomal enzyme, alpha-L-iduronidase treated with Aldurazyme® in home infusion setting according to authorized clinical practice and the approved risk management plan document (Cohort B).
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | For at least 12 months starting from enrollment (day 0)
  Treatment emergent adverse events (TEAEs) are defined as any event which are not present prior to the initiation of the Enzyme replacement therapy (ERT) administration in homecare setting or any event already present that worsens in either intensity or frequency following initiation of ERT administration in home-care setting.
Number of participants with treatment-emergent adverse events (TEAEs) for each class of severity | For at least 12 months starting from enrollment (day 0)
  TEAEs are defined as any event which are not present prior to the initiation of the ERT administration in homecare setting or any event already present that worsens in either intensity or frequency following initiation of ERT administration in home-care setting. An adverse event grading scale of mild, moderate and severe is used for grading of adverse event severity.
Number of participants with serious treatment-emergent adverse events (TEAEs) | For at least 12 months starting from enrollment (day 0)
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose: 1) results in death or 2) is life-threatening or 3) requires inpatient hospitalization or prolongation of existing hospitalization or 4) results in persistent or significant disability/incapacity or 5) is a congenital anomaly/birth defect or 6) is a medically important event.
Number of participants with treatment-emergent adverse events (TEAEs) related to alglucosidase or laronidase | For at least 12 months starting from enrollment (day 0)
  TEAEs are defined as any event which are not present prior to the initiation of the ERT administration in homecare setting or any event already present that worsens in either intensity or frequency following initiation of ERT administration in home-care setting. A TEAE is defined as treatment-related if it has a reasonable possibility that the event is related to alglucosidase or laronidase.
Number of participants with infusion associated reactions (IARs) | For at least 12 months starting from enrollment (day 0)
  IARs are defined as AEs that occur during either the infusion or the observation period following the infusion which are deemed to be related or possibly related to Myozyme® and Aldurazyme®. At the discretion of the Investigator, AEs occurring after completion of the post-infusion observation period that are assessed as related may also be considered IARs.
Number of participants with concomitant medications for each Anatomical Therapeutic Chemical (ATC) classification systems | At enrollment (day 0)
  Participants will be asked about their use of concomitant medication at enrollment.
Number of participants with change in the use of concomitant medications in case of non-tolerated infusion | For at least 12 months starting from enrollment (day 0)
  Participants will be asked about their perception regarding any additional medications or treatments or any changes in regimen or dosages compared to their baseline (day 0) state. Any change in the therapy (increased therapy, decrease therapy, no change in therapy) during the study will be reported.

SECONDARY OUTCOMES:
Patient satisfaction | For at least 12 months starting from enrollment (day 0)
  Patient satisfaction data will be collected through a satisfaction questionnaire, including potential benefits in terms of stress, time and costs. The questionnaire aims to evaluate patient satisfaction about home infusion: 1) where do you prefer to receive ERT, home or hospital; 2) why (list of reasons); 3) how do you feel now; 4) if you are in home infusion, how do you rate your health than when you were treated in hospital.
Patient compliance | For at least 12 months starting from enrollment (day 0)
  Patient compliance is assessed as number of missed infusions versus planned and/or return to hospital setting (with reasons).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Italy, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org